CLINICAL TRIAL: NCT05284383
Title: Reducing Nocebo Effects on Pressure Pain: open-and Closed-label Counterconditioning and Extinction Compared
Brief Title: Reducing Nocebo Effects on Pressure Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University (Other)
Responsible Party: Principal Investigator, Andrea W.M Evers, PhD, Professor, Leiden University Medical Center
Organization: Leiden University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2020-02-04-A.W.M.Evers-V1-2085
Record Dates: First submitted 2022-02-17; First posted 2022-03-17 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Pain; Hyperalgesia
Keywords: Pressure pain; Nocebo effect; Conditioning; Counterconditioning
MeSH Terms: conditions — Pain; Hyperalgesia

STUDY DESIGN:
Masking Description: One of the groups is an open-label group, meaning there is no masking. For the other two groups, participants are not aware of group allocation, but as verbal suggestions are given regarding the device, they are not fully masked (despite being unaware of the procedures that are used).
  Investigators are masked until the end of calibration, to prevent the influence of the investigator on the calibration process as much as possible. Afterwards, blinding of the investigator is not possible due to the nature of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Open-label counterconditioning (Experimental): Closed-label conditioning followed by open-label counterconditioning, using moderately painful stimuli (during conditioning) and non-painful stimuli (during counterconditioning), combined with closed-label nocebo suggestions and open-label nocebo reduction suggestions
  Interventions: Behavioral: Closed-label nocebo conditioning; Behavioral: Open-label counterconditioning
- Closed-label counterconditioning (Experimental): Closed-label conditioning followed by closed-label counterconditioning, using moderately painful stimuli (during conditioning) and non-painful stimuli (during counterconditioning), combined with closed-label nocebo suggestions and closed-label nocebo reduction suggestions
  Interventions: Behavioral: Closed-label nocebo conditioning; Behavioral: Closed-label counterconditioning
- Closed-label extinction (Active Comparator): Closed-label conditioning followed by closed-label extinction, using moderately painful stimuli (during conditioning) and slightly-painful stimuli (during extinction), combined with closed-label nocebo suggestions during conditioning and no/neutral suggestions during extinction
  Interventions: Behavioral: Closed-label nocebo conditioning; Behavioral: Closed-label extinction

INTERVENTIONS:
Behavioral: Closed-label nocebo conditioning — Conditioning consists of a learning and test phase. In the learning phase, a message indicating the sham activation of a Transcutaneous Electrical Nerve Stimulation (TENS) device (CS) will be repeatedly paired with a moderate intensity pressure pain stimulus, whereas a message indicating the deactivation of the sham device will be repeatedly paired with a slightly painful pressure pain stimulus. Participants will be given a verbal suggestion in line with the conditioning procedure (i.e. activation of the device will increase their pain). The testing phase is similar to the learning phase, but a slight pressure pain intensity is used for all trials, to test for a nocebo effect (i.e. to test whether participants score "TENS on" trials as more painful than "TENS off" trials).
Behavioral: Closed-label counterconditioning — Counterconditioning consists of a learning and test phase. In the learning phase, a message indicating the sham activation of the TENS device (CS) is now repeatedly paired with a non-painful intensity pressure pain stimulus, whereas a message indicating the sham deactivation of the TENS device will be repeatedly paired with a slightly painful pressure pain stimulus. Participants will be given a verbal suggestion in line with the counterconditioning procedure (i.e. activation of the device will reduce their pain). The testing phase is similar to the learning phase, but a slight pressure pain intensity is used for all trials, to test whether the nocebo effect is successfully reduced (i.e. to test whether participants no longer score "TENS on" trials as more painful than "TENS off" trials or even score "TENS on" trials as less painful).
  Arms: Closed-label counterconditioning
Behavioral: Open-label counterconditioning — Counterconditioning consists of a learning and test phase. In the learning phase, a message indicating the sham activation of the TENS device (CS) is now repeatedly paired with a non-painful intensity pressure pain stimulus, whereas a message indicating the sham deactivation of the TENS device will be repeatedly paired with a slightly painful pressure pain stimulus. Participants will be given a open-label verbal suggestions in line with the counterconditioning procedure (i.e. they are told counterconditioning will be used to reduce nocebo effects and they are told the device is sham, but that their pain will still be influenced because of the placebo effect). The testing phase is similar to the learning phase, but a slight pressure pain intensity is used for all trials, to test whether the nocebo effect is successfully reduced (i.e. to test whether participants no longer score "TENS on" trials as more painful than "TENS off" trials or even score "TENS on" trials as less painful).
  Arms: Open-label counterconditioning
Behavioral: Closed-label extinction — Extinction consists of a learning and test phase. In the learning phase, slightly painful stimuli are used for all trials. During the testing phase, again a slight pressure pain intensity is used for all trials, to test whether the nocebo effect is successfully reduced (i.e. to test whether participants no longer score "TENS on" trials as more painful than "TENS off" trials).
  Arms: Closed-label extinction

SUMMARY:
Nocebo effects are known to adversely affect the experience of various physical symptoms, such as pain and itch. Nocebo effects can be induced by associative learning mechanisms of classical conditioning. Furthermore, recent studies have shown that counterconditioning can successfully reduce nocebo effects, and to a larger extent than mere extinction, which suggests counterconditioning can be an innovative method for desensitization of symptoms. When using such procedures in clinical practice, deception of patients should be avoided as much as possible. The use of open-label procedures could provide a promising alternative. While previous studies have already shown that open-label placebos are effective, the effects of open-label counterconditioning and closed-label counterconditioning are not extensively investigated in comparison to other strategies, such as extinction, and not yet compared amongst each other. Before implementing such a procedure in clinical practice, it would be relevant to get an insight in the efficacy of both open- and closed-label counterconditioning in healthy participants as compared to extinction and to investigate whether open-label counterconditioning can be equally effective as closed-label counterconditioning. Furthermore, it would be relevant to study the induction and reduction of nocebo effects using a pain modality that mimics the type of pain that people suffering from several chronic pain conditions experience, such as pressure pain. The main aim of the current study is to investigate whether open- and closed-label counterconditioning are more effective in reducing nocebo effects than extinction. To this aim, it will be investigated whether open- and closed-label counterconditioning lead to stronger reductions in nocebo effects on pressure pain than (closed-label) extinction, and whether all three successfully reduce nocebo effects. Finally, it will be tested whether open- and closed label counterconditioning are comparable in effectivity.

DETAILED DESCRIPTION:
The primary objective of the study is to investigate whether open- and closed-label counterconditioning are more effective in reducing nocebo effects than extinction.

The experimental (open- and closed-label counterconditioning) and control (extinction) groups will be compared on the change in the nocebo effect from before to after counterconditioning. The nocebo effect is defined as the mean difference in self-reported pain ratings (on a numeric rating scale from 0 (no pain) to 10 (worst pain imaginable))during all experimental trials and control trials in the test phase of nocebo conditioning and the test phase of counterconditioning/extinction. The reduction of the nocebo effect will be determined by calculating the mean difference between the nocebo effect after conditioning and after counterconditioning/extinction. It is expected that participants in both counterconditioning groups will show a larger reduction of the nocebo effect than participants in the extinction group. A one-way ANOVA will be conducted, to examine the main effect of group on the amount of change in nocebo effects. Then, post-hoc analyses will be conducted after the primary analysis, to test for differences between the three forms of nocebo reduction.

Secondary, it will be tested whether all three procedures (open- and closed-label counterconditioning and extinction) lead to a significant reduction of the nocebo effect, by comparing the amount of reduction to test value 0. It is hypothesized that all groups show a significant reduction.

Finally, it will be investigated whether open- and closed-label counterconditioning procedures are comparable in terms of their ability to reduce nocebo effects on pressure pain. Both groups are expected to be comparable in efficacy of reducing the nocebo effect.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-35 years
* Good understanding of written and spoken Dutch or English

Exclusion Criteria:

* Severe somatic or psychiatric morbidity (e.g., heart/lung diseases, DSM-V psychiatric disorders)
* Raynaud's disease, chronic pain complaints at present or in the past
* Current pain complaints (> 2 on NRS)
* Current use of medication (except for birth-control pill)
* Injuries on the non-dominant hand
* Refusal/inability to remove nail polish or artificial nails for the experiment
* Pregnancy or breastfeeding

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2022-04-05 (Actual); Study Completion 2022-04-05 (Actual)

PRIMARY OUTCOMES:
Nocebo reduction; group comparison | On the testing day; testing phase of nocebo induction and reduction
  The change in nocebo effects from after nocebo conditioning (part 1) to after either form of counterconditioning or extinction (part 2) will be compared between groups. The nocebo effect is defined as the difference between the pain scored during experimental trials (on a 0-10 NRS) and during control trials (same NRS). The change is calculated by subtracting the nocebo effect after counterconditioning from the nocebo effect after nocebo conditioning.

SECONDARY OUTCOMES:
Nocebo reduction | On the testing day; testing phase of nocebo induction and reduction
  For all three groups separately, it will be tested whether the nocebo effect is significantly reduced from test phase of nocebo conditioning to the test phase of either form of counterconditioning or extinction. The nocebo effect is defined as the difference between the pain scored during experimental trials (on a 0-10 NRS) and during control trials (same NRS). Nocebo reduction is calculated by subtracting the nocebo effect after counterconditioning from the nocebo effect after nocebo conditioning. For all groups separately, the amount of reduction will be compared to test value 0.
Nocebo reduction; equivalence of the two forms of counterconditioning | On the testing day; testing phase of nocebo induction and reduction
  It will be tested whether the change in nocebo effects from the test phase of conditioning to the test phase of counterconditioning in the open- and closed-label groups is comparable. The nocebo effect is defined as the difference between the pain scored during experimental trials (on 0-10 NRS) and during control trials (same NRS). The change is calculated by subtracting the nocebo effects after counterconditioning from the nocebo effect after nocebo conditioning.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Evers, Prof, Principal Investigator — Leiden University
Locations (1):
- Leiden University, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
All data are collected pseudonymised; consent forms are the only sources containing personal data and will not be shared, but are monitored by the department's Data Monitor.
Supporting Information: SAP, Analytic Code
Time Frame: Data will become available immediately after study publication and will be retained for 15 years.
Access Criteria: Data can be shared with scientists in relevant fields for the purpose of future studies such as replication or meta-analysis (or with designated persons for monitoring purposes).